CLINICAL TRIAL: NCT04239950
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Placebo Controlled Study to Evaluate the Efficacy and Safety of Ethyl Icosapentate in Patients With Severe Hypertriglyceridemia
Brief Title: Efficacy of Ethyl Icosapentate in Patients With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MND2112H33; 20191474 (Registry Identifier: ChiCTR)
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — eicosapentaenoic acid ethanolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, orally, twice daily after breakfast and dinner for 12 weeks.
  Interventions: Drug: Placebo
- Ethyl Icosapentate 1.8g (Experimental): Ethyl Icosapentate 0.9g, orally, twice daily after breakfast and dinner for 12 weeks.
  Interventions: Drug: Ethyl Icosapentate
- Ethyl Icosapentate 3.6g (Experimental): Ethyl Icosapentate 1.8g, orally, twice daily after breakfast and dinner for 12 weeks.
  Interventions: Drug: Ethyl Icosapentate

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Ethyl Icosapentate — Ethyl Icosapentate
  Arms: Ethyl Icosapentate 1.8g; Ethyl Icosapentate 3.6g

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ethyl icosapentate in Chinese patients with severe hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria

1. Patients whose serum Triglyceride (TG) level (fasting) from week -6 to week -4 is 500 mg/dL or higher and less than 2,000 mg/dL
2. Patients who receive instructions for lifestyle improvement and are able to comply with all instructions throughout the study participation period
3. Patients who are 18 to < 75 years of age, regardless of sex, at the time of informed consent
4. Patients who have provided written consent to participate in this clinical trial
5. Patients whose serum TG level (fasting) is less than 2,000 mg/dL at Week -2
6. Patients whose serum TG level (fasting) is less than 2,000 mg/dL at Week -1
7. Patients in whom the average of Week -2 and Week -1 in serum TG level (fasting) is 500 mg/dL or higher and less than 2,000 mg/dL
8. Outpatients

Exclusion Criteria:

1. Patients whose HbA1c from week -6 to week -4 is 8.0% or higher
2. Patients whose Alanine Aminotransferase (ALT) or Aspartate aminotransferase (AST) from week -6 to week -4 is more than 3 times the upper limit of normal
3. Patients with, or with a history of, angina pectoris or myocardial infarction
4. Patients with a history of percutaneous transluminal coronary angioplasty or coronary artery bypass grafting
5. Patients with familial lipoprotein lipase (LPL) deficiency, familial apolipoprotein C-II (apo C-II) deficiency, or familial type III, IV hyperlipidemia
6. Patients with hypothyroidism, Cushing's syndrome, acromegaly, nephrotic syndrome, chronic renal failure, systemic lupus erythematosus, myeloma, or nonalcoholic steatohepatitis (NASH)
7. Patients with hyperlipidemia induced by drugs (e.g., corticosteroids, beta-blockers, contraceptives, interferons, retinoids, and diuretics)
8. Patients with, or with a history of, alcohol dependence or abuse or patients whose hyperlipidemia is presumed to be primarily caused by alcohol
9. Patients with aortic aneurysm or who have undergone aortic aneurysmectomy within the last 6 months
10. Patients with uncontrollable hypertension (patients with a systolic blood pressure of ≥180 mmHg or a diastolic blood pressure of ≥110 mmHg in a sitting position at Visit 1 (Week -4))
11. Patients with, or with a history of, pancreatitis or patients suspected as pancreatitis by examination, etc
12. Patients with a diagnosis of complication of pancreas or bile duct-related neoplastic disease
13. Patients with type 1 diabetes mellitus or type 2 diabetes mellitus requiring insulin therapy
14. Patients with any of the following hemorrhagic findings within the last 6 months:

    * Patients with, or with a history of, clinically significant hemorrhagic disease (e.g., cerebral hemorrhage, hemophilia, capillary fragility, gastrointestinal [GI] ulcer, urinary tract hemorrhage, hemoptysis, vitreous hemorrhage)
    * Patients with clinically significant bleeding tendency (e.g., menorrhagia, frequent epistaxis)
    * Patients with, or with a history of, severe trauma
    * Patients with a history of surgery requiring blood transfusion
15. Patients who have taken any EPA product
16. Patients who have received a PCSK9 (human proprotein convertase subtilisin/kexin type 9) inhibitor to treat hyperlipidemia
17. Patients who have taken antihyperlipidemic drugs within the last 4 weeks
18. Pregnant, possibly pregnant, or lactating women
19. Patients with a history of hypersensitivity to polyunsaturated fatty acids or gelatin
20. Patients with, or with a history of, malignant tumor
21. Patients with any serious disease, including hepatic, renal, hematologic, respiratory, GI, cardiovascular, psychological, neurologic, metabolic, and electrolyte disorders, or hypersensitivity
22. Patients who have received any other investigational drug within the last 3 months
23. Patients who are judged by the principal (or sub-) investigator to be ineligible as a study subject for any other reason
24. Patients with a systolic blood pressure of ≥180 mmHg or a diastolic blood pressure of ≥110 mmHg at Visit 2 (Week -2))
25. Patients who have changed the dosage of antidiabetic drug (except insulin) or who have switched from one drug to another since Visit 1 (Week -4)
26. Patients with a systolic blood pressure of ≥180 mmHg or a diastolic blood pressure of ≥110 mmHg at Visit 3 (Week -1)
27. Patients with an HbA1c level of ≥8.0% at Visit 2 (Week -2)
28. Patients whose ALT or AST is more than 3 times the upper limit of normal at Visit 2 (Week -2)
29. Patients with a systolic blood pressure of ≥180 mmHg or a diastolic blood pressure of ≥110 mmHg at Visit 4 (Week 0)
30. Patients with an HbA1c level of ≥8.0% at Visit 3 (Week -1)
31. Patients whose ALT or AST is more than 3 times the upper limit of normal at Visit 3 (Week -1)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2020-05-09 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Percentage of change from baseline in serum triglyceride level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Adverse events after the start of study drug administration | 12 weeks

SECONDARY OUTCOMES:
Percentage of change from baseline in serum total cholesterol level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum low-density lipoprotein cholesterol (LDL-C) level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Percentage of change from baseline in serum high-density lipoprotein cholesterol (HDL-C) level at 12 weeks after the start of study drug administration | Baseline and 12 weeks
Adverse drug reaction after the start of study drug administration | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takuya Mori, Study Director — Mochida Pharmaceutical Company, Ltd.
Locations (1):
- Mochida Investigational sites, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Long M, Chen F, Wu D, Pei Z, Wang X, Zhao W, Mori T, Zhao S. Efficacy and safety of highly purified ethyl icosapentate soft capsules (MND-21) for the treatment of severe hypertriglyceridemia: A 12-week, multi-center, placebo-controlled, randomized, double-blind, phase III clinical trial in China. J Clin Lipidol. 2025 Dec 14:S1933-2874(25)00539-2. doi: 10.1016/j.jacl.2025.12.007. Online ahead of print. PMID 41500861